CLINICAL TRIAL: NCT04251468
Title: Clinical Potassium Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: NGFI Next Generation Fluorescence Imaging GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CPPS
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Hyperkalemia
Keywords: plasma potassium measurement; saliva potassium measurement; hemodialysis; fluorescence assay; ECG-based potassium estimation; Förster resonance energy transfer
MeSH Terms: conditions — Hyperkalemia | interventions — Ion-Selective Electrodes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEPII (Other): All patients who completed the study.
  Interventions: Device: GEPII; Device: Ion-selective electrodes

INTERVENTIONS:
Device: GEPII — Saliva probes (K+Sa) will be measured using genetically encoded potassium ion indicators (GEPIIs)
Device: Ion-selective electrodes — Plasma potassium levels (K+Pl) will be measured using standard ion-selective electrodes.

SUMMARY:
In this pilot study, 30 prevalent hemodialysis patients will undergo three regular hemodialysis sessions during which various potassium assessments will be performed. Pre- (t1) and post-dialysis (t2) plasma potassium levels (K+Pl) will be measured using standard ion-selective electrodes. These values will be correlated to K+ determine in saliva probes (K+Sa) using genetically encoded potassium ion indicators (GEPIIs). Additionally, continuous ECG will be recorded during each hemodialysis treatment and potassium assessment (K+ECG) will be performed upon ECG-based parameters and correlated to K+Pl.

DETAILED DESCRIPTION:
Cardiovascular diseases are among the leading causes of death in industrialized countries. Medical therapy for these diseases has seen significant progress, much of which is based on agents interfering with the renin-angiotensin-aldosterone system (angiotensin-converting enzyme inhibitors, angiotensin receptor antagonists, mineralocorticoid receptor antagonists, neprilysin inhibitors). However, these agents bear the side effect of reducing renal potassium (K+) excretion and may thus lead to elevation of blood K+ Levels (hyperkalemia). Hyperkalemia is a potentially life-threatening condition, which in its most severe forms requires immediate medical attention, since there is imminent danger of dangerous arrhythmias and sudden cardiac death. Therefore, hyperkalemia is a leading reason to withdraw potentially lifesaving therapy in a significant number of patients, which is considered to have a negative impact on patient outcomes. Recently, novel intestinal potassium binders have been shown to be efficient in reducing incidence and severity of hyperkalemia These compounds have very recently been shown to allow extending the benefits of antihypertensive therapy with spironolactone to patients with chronic kidney disease with refractory hypertension . Yet due to preanalytical problems as well as time and cost-restraints, out-patient monitoring of serum or plasma potassium levels has proven problematic.

The plasma potassium level and kinetics at two timepoints before and after a hemodialysis session as determined by either standard of care (i.e. ion selective electrode) will be compared to the potassium level measured in (i) saliva (salivary potassium [K+Sa]) or (ii) determined based on electrocardiogram (K+ECG). Patients suffering from end-stage renal disease undergoing hemodialysis (HD) frequently present with severe hyperkalemia prior to a HD session. During HD treatment, K+ levels undergo unphysiologically rapid changes due to K+ removal via HD as well as due to changes in acid-base status. Thus, HD patients represent a unique population in whom significant K+ derangements and rapid K+ Level changes predictably occur and where these phenomena can be investigated in a safe environment.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 90 years of age
* End stage-renal disease or acute kidney injury patient undergoing hemodialysis
* Ability to provide oral and written informed consent
* Ability and willingness to comply with study procedures
* Willingness to not consume foods or drinks other than water during dialysis session

Exclusion Criteria:

* Intraventricular conduction abnormalities (left- or right bundle branch block, trifascicular block) which interfere with K+ECG determination
* Active inflammation or infection of the oral mucous membranes or dentition

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Relative difference in change of K+Sa at t2 versus t1 | Pre- (t1) and immediately post-dialysis (t2)
  Assess the performance of K+Sa compared to K+Pl
ECG P wave height | Pre- (t1) and immediately post-dialysis (t2)
  Comparison of the relative change of K+ECG at t2 versus t1
ECG PR interval | Pre- (t1) and immediately post-dialysis (t2)
  Comparison of the relative change of K+ECG at t2 versus t1
ECG QRS duration | Pre- (t1) and immediately post-dialysis (t2)
  Comparison of the relative change of K+ECG at t2 versus t1
ECG maximum R wave height | Pre- (t1) and immediately post-dialysis (t2)
  Comparison of the relative change of K+ECG at t2 versus t1
ECG QT interval | Pre- (t1) and immediately post-dialysis (t2)
  Comparison of the relative change of K+ECG at t2 versus t1
ECG ST segment depression | Pre- (t1) and immediately post-dialysis (t2)
  Comparison of the relative change of K+ECG at t2 versus t1
ECG maximum T wave height | Pre- (t1) and immediately post-dialysis (t2)
  Comparison of the relative change of K+ECG at t2 versus t1

SECONDARY OUTCOMES:
Percentage of false positive measurements, i.e. percentage where severe hyperkalemia [K+>6.0 mmol/L] was detected by means of K+ECG, which was not present in K+Pl | Pre- (t1) and immediately post-dialysis (t2)
  Assess the performance of K+ECG compared to K+Pl
Percentage of false negative measurement, i.e. percentage where severe hyperkalemia [K+>6.0 mmol/L] was not detected by means of K+ECG, which was present in K+Pl | Pre- (t1) and immediately post-dialysis (t2)
  Assess the performance of K+ECG compared to K+Pl
Severe hyperkalemia [K+Pl ≥ 6.5 mmol/L] detection rate using K+ECG: comparison of automated detection using the K+ECG algorithm vs experienced electrophysiologist. | Pre- (t1) and immediately post-dialysis (t2)
  Assess the performance of K+ECG algorithm vs experienced electrophysiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander H. Kirsch, MD, Principal Investigator — Medical University of Graz; Andras T. Deak, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No